CLINICAL TRIAL: NCT04564404
Title: Neuromusculaire Monitoring Survey - Financial
Brief Title: Neuromusculaire Monitoring Survey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EUNeuroMuscMonitoringSurvey2
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-09

CONDITIONS: Survey, Financial
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Questionnaire to ask about the willingness-to-buy applications in neuromuscular monitoring.

SUMMARY:
This survey aims to better define the willingness-to-buy for Applications in Neuromuscular Monitoring throughout European hospitals.

DETAILED DESCRIPTION:
This study consists of a simple online survey that takes approximately 2 minutes to complete.

The study aims to assess the willingness-to-buy for Applications in Neuromuscular Monitoring (monitoring and software-based) within the anesthesia departments of European hospitals. The survey is targeted to the department heads of the questioned anesthesia departments.

ELIGIBILITY:
Inclusion Criteria:

* Active Anesthesiology department heads of European Anesthesiology departments.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Willingness to buy questionnaire | 4 months
  Would this person be willing to buy neuromuscular monitoring applications.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided